CLINICAL TRIAL: NCT04385784
Title: Effectiveness of a Postural Control Exercise Program on Balance and Risk of Falls in Sedentary Older Adults.
Brief Title: Postural Balance Program in Sedentary Older Adults.
Acronym: PEMaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Pérez-Robledo, Fátima, Professor (Associate), University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10.14201/gredos.140334
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Postural Balance
Keywords: Postural balance; Aged; Sedentary Behavior; Exercise Therapy
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The study is interventional, consisting of three arms with parallel monitoring. The first two arms perform an intervention based on physical exercise guided by physiotherapists, in order to improve their balance and postural control. These two arms are differentiated by the level of daily physical activity that their participants have (sedentary and active people). In addition to the guided exercise sessions, they are offered an exercise book to perform at home. The third arm of the study only performs the home-based program and is made up of sedentary people.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sedentary Intervention Group (SIG) (Experimental): Group of sedentary older adults who perform the intervention and a home-based exercise program.
  Interventions: Other: Balance exercise program.; Other: Home-based exercise program.
- Active Intervention Group (AIG) (Experimental): Group of active older adults who perform the intervention and a home-based exercise program.
  Interventions: Other: Balance exercise program.; Other: Home-based exercise program.
- Control Group (CG) (Active Comparator): Group of sedentary older adults who perform a home-based exercise program.
  Interventions: Other: Home-based exercise program.

INTERVENTIONS:
Other: Balance exercise program. — Multimodal exercise program that combines strength, mobility, elasticity and postural control exercises. It develops once a week for a total of 24 weeks. Each session lasts one hour and is carried out in small groups of 8 to 10 people maximum.
  Arms: Active Intervention Group (AIG); Sedentary Intervention Group (SIG)
Other: Home-based exercise program. — Exercises based on the OTAGO program that are carried out at home without supervision. Participants are explained to carry out the program three or four times a week in a safely way.

SUMMARY:
Introduction: Balance is one of the physical capacities that are altered due to the changes produced by aging. This represents an increased risk of falls in older adults. In Spain, the percentage of older people who fall each year is high and carries a series of important economic and social consequences. Sedentary lifestyle complicates this process, further increasing the risk of falls in older adults.

Objective: To design and apply a postural control exercise program to improve balance and reduce the risk of falls in healthy sedentary older adults.

Material and methods: Longitudinal, prospective, quasi-experimental study, in which a balance program of one weekly session for 24 weeks was developed. 112 healthy people over 60 years of age participated and were randomly divided into three work groups: Active Intervention Group (GIA), Sedentary Intervention Group (GIS) and Control Group (CG). His steady state and risk of falls were analyzed with the following functional tests: Tinetti Scale, Timed Up & Go Timed Test (TUG), One-Legged Stance Test (OLS), Fullerton Advanced Balance Scale (FAB) and 30 Second Chair Stand Test (30SCST). The GIA and GIS carried out the balance program and received a workbook to carry out at home. The CG only performed the home exercises.

DETAILED DESCRIPTION:
INTERVENTION PROTOCOL The target population of our study were older people belonging to one of the older people's associations in the town of Salamanca. The program was offered in the different associations and an inscription sheet was passed in which they had to provide different information related to their personal situation. All the people he wanted signed up.

Once all the participants enrolled in the program, a draw of places was done to guarantee the randomization of the sample, assigning the participants to the intervention group or the control group.

To ensure a sample size with a confidence level of 95% and an error rate of 10%, a larger sample of 96 people was assumed. A total of 112 participants were included in the program.

An initial assessment was made of all program participants, regardless of the group to which they were assigned. In this session, they were given an informed consent that they had to sign it in order to participate in the program.

The most important data when selecting the elderly is the level of physical activity they carry out in their day to day. In this way, the elderly were divided into two groups: a trained group, that is, who was doing physical activity at the current time and had done it during the previous year, regardless of the type it was, according to the criteria established by WHO; and a sedentary group, which included those elderly who did not meet the minimum criteria for recommended physical activity.

Initial Assessment

The initial assessment was carried out during the first week of the intervention. All the participants did it regardless of the group to which they belonged. The following tests were carried out to evaluate the participants:

* Anthropometric analysis (weight, height, BMI).
* Fullerton Advanced Balance Scale.
* Tinetti Scale (balance and gait).
* Timed Up & Go Test.
* One-leg Stance test.
* 30 Second Chair Stand Test.

Intervention Groups Both the intervention group made up of active people (AIG) and the group made up of sedentary people (SIG), started the intervention after carrying out the initial assessment. To avoid bias, the participants and the physiotherapists in charge of giving the sessions were blinded without knowing the group to which they belonged. Only the principal investigator responsible for conducting the initial assessment knew about the division.

Participants developed the balance program for a total of 24 weeks. The sessions were performed once a week, lasting 55-60 minutes.

The sessions had an individual part and a group part, with a short break within them.. In addition to the exercise protocol as such, guidelines were taught to perform the home-based workbook in a safe and appropriate manner.

After this period, a final assessment was carried out, where all the participants were reviewed again.

Intervention

For the design of the standard session, warm-up exercises, muscle strength, postural control and stretching were included, in addition to dedicating time to hydration. Hydration is not considered exercise as such, but it is considered necessary during the session, since it is essential for older people. The plan used to design the sessions is detailed below:

1. Warm-up.
2. Muscle strength exercises.
3. Individual postural control exercises.
4. Hydration.
5. Groupal postural control exercises.
6. Stretching and ventilation exercises. It is recommended to wear comfortable and wide clothing that allows the necessary movements to be carried out and avoids friction and discomfort. The indicated shoes are comfortable sports shoes, avoiding high-heeled shoes, shoes that are too tight or shoes that do not fit well and produce imbalances.

Before starting the program, the participants were informed that they should try to carry out the exercises as correctly as possible, making an effort, but that each person should adapt the exercise to their level, carrying out the activity safely and avoiding dangers. In addition, the physiotherapists in charge of directing the activity, during the progression of the sessions indicated to the participants those variations that they considered necessary for the exercise to be safe but effective, progressing in the difficulty as the physical condition of the participant required it.

At the beginning of the session there was a greeting and a count of the participants, to control attendance and check the clothing of each one.

1. - Warm-up The warm-up always includes the same exercises, which allow the participants to become familiar with them and introduce the exercises of strength and postural control. This part of the session includes the first 10 minutes of it.
2. - Exercises of muscular strength These exercises are performed for approximately 10 minutes. The exercises are alternated throughout the sessions, in such a way that, each week, the upper or lower body is worked more.
3. - Individual postural control exercises The duration of this part of the session is approximately 10 minutes, alternating exercises throughout the program. During this part of the session, the physical therapists who lead the activity pay special attention to how the participants perform the exercises, correcting and giving the appropriate instructions when necessary.
4. - Hydration Each session is given a break of approximately 5 minutes to hydrate. In each session, participants are reminded to bring a bottle of water or juice to hydrate properly. Older adults are a risk group for dehydration. This can be aggravated during physical exercise. Therefore, it is recommended to hydrate during the sessions, to avoid problems associated with dehydration, such as urinary infections, constipation or hypotension.
5. - Groupal postural control exercises After hydration, the session is continued with postural control exercises, but including group activities so that there is a more playful part and, thus, increase the motivation of the participants.
6. - Stretching and ventilation exercises At the end of the previous activity, stretching exercises of the different muscle groups are carried out, as well as mobility exercises accompanied by respiratory movements to return to rest and lower heart rate. This part of the session lasts approximately 10 minutes.
7. - Precautions and exercises to avoid Exercises that keep the head below the level of the waist, which involve hyperflexion, hyperextension, or hyperrotation of the spine or other joints, should be avoided.

Exercises must be done safely and comfortably. Any exercise that causes discomfort or pain on the participants should be avoided.

All exercises must be carried out safely, if they require supports they must be stable and physiotherapists must ensure that no participant is in danger of falling..

Control Group The target population were older people who decided to enroll in the program voluntarily and who were sedentary, that is, who did not meet the WHO criteria of recommended physical activity for their age group.

The objective of having this control group was to determine the effectiveness of the program and the usefulness of having a professional who teaches and trains individuals. We wanted to see if the program improved the physical capacity of the participants and if the presence of a professional as well as attendance at a regular activity is beneficial and determines greater changes in the subjects' abilities.

The control group should be composed of sedentary people, since in previous studies it was seen that attendance at physical activity programs, such as the Geriatric Revitalization Program (PReGe) carried out by the University of Salamanca, determined sufficient changes to improve the balance of participants.

The group consisted of those participants who during the draw were not selected for the intervention group. Not all of them formed the group but after the initial assessment and determine the level of physical activity each were selected those who were sedentary, and those who were active were excluded from the study.

During the assessment session, they were also given a notebook where some exercises to improve balance were explained in detail and they were instructed to do them at least twice a week.

After 24 weeks, they were asked to pass the assessment tests again and thus it was determined whether the indication of home-base exercise had any effect on the physical abilities of the subjects.

Final Assessment At the end of the intervention period, a final assessment was carried out by both groups, which included the same tests as the initial assessment.

Statistical analysis of the data For the storage, treatment and statistical analysis of the data, the statistical package IBM-SPSS-Statistics, version 23.0, for Windows was used.

The data was digitized and, afterwards, an exhaustive descriptive analysis of all the variables was performed to detect possible errors in the collection or digitization of the data, mainly affecting the maximum and minimum of the quantitative variables.

Once the definitive data matrix was defined, a descriptive analysis of the different variables and data collected during the initial assessment was carried out, as well as an analysis of data by protocol. To determine which statistic corresponds to them, firstly, a normality test of each variable was performed with the Shapiro-Wilk Test, one of the most powerful tests, especially with small samples, as is our case.

In the event that the variable followed a normal distribution, the mean (M) and standard deviation (DT) were calculated. If the variable did not follow the normal distribution, the median and interquartile range were calculated. In the case of categorical variables, the results were expressed in percentages.

The descriptive study was carried out, segmenting the sample and dividing it by sex, age, activity level and BMI.

In the descriptive analysis of the variables related to balance and the risk of falls, the percentage of people who were at risk of falls was calculated for each of the variables.

For the comparative analysis between two quantitative variables, the T-Student test was used, if the variables behaved normally, and the U-Mann-Withney test when any of the variables did not follow a normal distribution.

In the case of categorical or qualitative variables, they used contingency tables and the Chi-square test to analyze the results obtained.

For the inferential analysis of the data, whenever there were more than two variables for the analysis, the F-Snedecor test (ANOVA) was performed if the variables were normal, or the H-Kruskal-Wallis test, when any of the variables were not maintained a normal distribution.

Contrast tests were performed, in the event that there were significant differences in the tests of multiple variables. To determine between which groups there were differences, t tests were used to determine the contrast.

The calculation of correlations was also performed, using the Pearson's correlation coefficient, for quantitative variables, or the Spearman correlation coefficient, in the event that any of the variables was categorical.

In all analyzes, a 95% confidence interval was established with significance indices of p <0.05. The results obtained have been expressed with the value of the statistician, as well as the p-values and those data that are most interesting for the interpretation of the results.

ELIGIBILITY:
Inclusion Criteria:

* People over 60 year who decide to participate voluntarily.
* Attendance at the Initial Assessment.
* Acceptance of Informed Consent.

Exclusion Criteria:

* Presence of absolute or relative contraindications to physical exercise.
* Presence of serious balance limitations, such as severe neurological, visual or musculoskeletal disorders.
* Presence of difficulties to carry out the tests of the Initial Assessment.
* Incidents or pathologies suffered during the intervention that interfere with the study.
* Failure to attend the Final Assessment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Weekly physical activity | 1 year
  The number of hours and the intensity level of the physical activity carried out by the participants habitually are recorded. Thus, according to the criteria established by WHO, physically active people are differentiated from sedentary people. It is a variable that determines the group in which the participants are included.
Fullerton Advanced Balance Scale (FAB) | 24 weeks
  It is a validated balance measurement scale in older adults. It consists of 14 items that assess different aspects of the static and dynamic balance. Each item scores from 0 to 4 points, and a total score of 56 points can be achieved. A score below 25 points indicates a high risk of falls.
Tinetti Scale | 24 weeks
  It is a validated scale to assess the risk of falls in older adults. It consists of two sections, the first is gait with 12 possible points, and the other is balance with 16 possible points. The maximum score that can be achieved is 28 points. A score below 19 points indicates high risk of falls.
Test Timed Up & Go (TUG) | 24 weeks
  It is a validated test to determine the functionality and risk of falls in older adults. To assess it, the time it takes for a person to get up from a chair, walk 6 meters and sit is timed. A score below 10 seconds indicates a high risk of falling.
One-Leg Stance Test (OLS) | 24 weeks
  This test evaluates the static balance and the risk of falls of older adults. It consists of maintaining the position on one leg as long as possible. A maximum time of 30 seconds is established. It is done with both legs. A person who holds the position for less than 10 seconds is at risk of falling.
30 Second Chair Stand Test (30SCST) | 24 weeks
  This test is validated to measure strength in the lower extremities as well as the risk of falls in older adults. It consists of counting the number of times a person can stand up and sit down in 30 seconds. There are normal values for each age and sex with which the participant is assess.
Number of Falls | 24 weeks
  The number of falls suffered by the participant during the last 6 months is recorded.

SECONDARY OUTCOMES:
Sex | 24 weeks
  The sex of the participants is recorded at the start of the study.
Date of birth | 24 weeks
  The participant's date of birth is collected in order to calculate his age in years.
Weight | 24 weeks
  The weight of the participants is analyzed in kilograms.
Height | 24 weeks
  The height of the subject is determined in meters.
Body Mass Index (BMI) | 24 weeks
  The participant's BMI is calculated from his height and weight.
Adherence | 24 weeks
  Adherence to the program is calculated from the record of the percentage of attendance at the intervention sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No